CLINICAL TRIAL: NCT00131014
Title: Establishing a Tumor Bank and Initial Analysis of Germline and Tumor-Related Genetic Alterations in Families With Multiple Lymphoproliferative Malignancies
Brief Title: Establishing a Tumor Bank in Families With Multiple Lymphoproliferative Malignancies
Status: Recruiting | Type: Observational
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Jennifer R. Brown, MD, PhD, Assistant Professor of Medicine, Dana-Farber Cancer Institute
Other Study IDs: 04-165
Record Dates: First submitted 2005-08-15; First posted 2005-08-17 (Estimated); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Non-Hodgkin's Lymphoma; Hodgkin's Disease; Leukemia, Lymphocytic, Chronic; Lymphoproliferative Disorders
Keywords: Non-Hodgkin's Lymphoma; Hodgkin's disease; Chronic Lymphocytic Leukemia; Lymphoproliferative disorder; Genetics
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Hodgkin Disease; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoproliferative Disorders

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood Cheek cells Paraffin blocks of tumor tissue

GROUPS / COHORTS (3):
- Next of Kin of deceased subj by lymphoma: Next of Kin of deceased subject by lymphoma
- Subject unaffected by lymphoma: Subject unaffected by lymphoma
- Subject affected by lymphoma: Subject affected by lymphoma

SUMMARY:
The purpose of this study is to investigate possible genetic factors that contribute to the development of lymphomas. The databank will be used to determine whether familial lymphomas have unique genetic characteristics different from sporadic lymphomas and to attempt to identify a gene that confers an increased risk of lymphoma.

DETAILED DESCRIPTION:
* Patients who participate will be asked to complete detailed family and medical history questionnaires initially, with a follow-up questionnaire every year.
* Patients will be asked to supply a blood sample and possibly a mouthwash sample, both of which can be done by mail.
* Patients will be asked to consent to the release of their lymphoma tissue block for the purposes of the study.
* Patients will be given letters of invitation for their affected relatives to invite them to participate.

ELIGIBILITY:
Inclusion Criteria:

* Any individual diagnosed with non-Hodgkin's lymphoma or Hodgkin's disease or chronic lymphocytic leukemia (CLL), who has a 1st degree relative (parent, sibling or child) with a lymphoproliferative disorder; or families in which the individual has a lymphoproliferative disorder, and an unusual clustering of frequent or premature solid tumors is also observed.
* Family members of the individual, either affected or unaffected with lymphoma, who are contacted by the individual and agree to participate in the study.
* Deceased family members may be included in the study. Public records such as death certificates may be used to confirm the history. Consent for medical records or tissue blocks will be obtained from the deceased family member's next of kin. The hierarchy of relatives defined as next of kin is spouse, offspring, parents and siblings. Archived tissue samples may be used for genetic research.
* Age > 18 years

Exclusion Criteria:

* Subjects without a family history of lymphoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Group 1: Next of kin of a relative who has died from lymphoma Group 2: Subjects who have a next of kin diagnosed with lymphoma and/or CLL Group 3: Subjects who have had or have non-Hodgkin's lymphoma, CLL or Hodgkin's disease and had a relative who also had lymphoma or CLL
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2004-08-09 (Actual); Primary Completion 2033-01 (Estimated); Study Completion 2033-01 (Estimated)

PRIMARY OUTCOMES:
Genetic factors that contribute to the development of lymphomas and CLL | Indefinite
  Genetic factors that contribute to the development of lymphomas and CLL

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer R. Brown, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States